CLINICAL TRIAL: NCT02263703
Title: Immunogenicity and Duration of Immunity in Immunosuppressed Children Vaccinated With Quadrivalent HPV Vaccine
Brief Title: Immunogenicity of HPV Vaccine in Immunosuppressed Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: Sydney Children's Hospitals Network (Other); Women's and Children's Hospital, Australia (Other Government)
Responsible Party: Principal Investigator, Prof Raina MacIntyre, Head of School and Professor of Infectious Diseases Epidemiology, The University of New South Wales
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007/028
Record Dates: First submitted 2014-10-03; First posted 2014-10-13 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Autoimmune Disease; Juvenile Idiopathic Arthritis; Inflammatory Bowel Disease; Evidence of Liver Transplantation; Kidney Transplant Infection; Bone Marrow Transplant Infection
Keywords: HPV vaccine, children, immunocompromised
MeSH Terms: conditions — Autoimmune Diseases; Arthritis, Juvenile; Inflammatory Bowel Diseases | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HPV vaccine (Experimental): Quadrivalent HPV vaccine
  Interventions: Biological: Quadrivalent HPV vaccine

INTERVENTIONS:
Biological: Quadrivalent HPV vaccine — Three 0.5 mL doses will be given at time 0, 2 months after the 1st dose and then 6 months after the initial dose. For kidney transplant recipients the first dose will be at least 6 months post-transplant.

SUMMARY:
Genital HPV is the necessary cause for cervical cancer, as well as a major contributing cause of several other cancers and conditions. There are now effective vaccines against the main oncogenic HPV types, HPV16 and 18.

Most research and discussion has focused on targeting the vaccine to young women and older adolescents. Based on this, a national free HPV vaccination program for adolescent girls commenced in 2007, in Australia. However, at the time of commencement, there had been no research on the use of this vaccine in immunosuppressed. Therefore, information on the immunogenicity, safety and duration of efficacy of HPV vaccine when administered to immunosuppressed children is needed. This trial looked at a 3 dose schedule of quadrivalent HPV vaccine in a range of immunosuppressed children, with the endpoint being immunogenicity, followed for 5 years for duration of immunity.

DETAILED DESCRIPTION:
To determine the immunogenicity, safety and persistence of immunity following human papillomavirus (HPV) vaccination in three groups of immunosuppressed children: recipients of allogenic bone marrow transplant, recipients of renal and liver transplants, and patients with juvenile chronic arthritis, inflammatory bowel disease and other autoimmune conditions who are on longterm immunosuppressive therapy.

Significance: Immunosuppressed populations are diverse in terms of degree, type and duration of immunosuppression. The study compares several groups in order to address the heterogeneity of immunosuppression and how this affects vaccine response. BMT patients have extreme, severe immunosuppression in the short term, but recover immune function with time. In contrast, solid organ transplant recipients have ongoing, chronic immunosuppression. Although successful cessation of immunosuppressives in liver transplant patients has been reported, most patients require ongoing treatment. The inflammatory bowel disease group of patients represents a non-transplant group who require ongoing, often low level immunosuppression, often with corticosteroids. Our study will compare these three groups, followed up for five years for duration of immunity. Time of vaccines, time of serological measures of immune response are as follows.

Serum collections:

0 - Baseline (before HPV vaccine dose 1); 2 months - At the time of receipt of HPV vaccine dose 2 (to measure response to dose 1); 6 months - At the time of receipt of HPV vaccine dose 3 (to measure response to dose 2); 7 months - 1 month after HPV vaccine dose 3; 12 months - after HPV vaccine dose 1; 2 years after HPV vaccine dose 1; 3 years after HPV vaccine dose 1; 4 years after HPV vaccine dose 1; 5 years after HPV vaccine dose 1.

ELIGIBILITY:
Inclusion Criteria:

- Immunosuppressed patients with following diseases; Bone marrow transplant recipients, liver transplant patients, renal transplant, Children with inflammatory bowel disease, juvenile Idiopathic arthritis and autoimmune conditions.

Exclusion Criteria:

* A platelet count of <50
* Immunoglobulin therapy within 3 months.
* Yeast allergy
* Any other known allergies to one of the vaccine component

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 2 years
  Indicator:
  1. Geometric mean four fold rises (with 95% confidence intervals) of the vaccine serotype specific IgG antibody in all participants.
  2. Proportion of subjects achieving a 4 fold rise in antibody titre for each serotype. Serum antibody levels will be measured using a Luminex immunoassay.
  Analysis: For each individual, the change in log-22FA levels for each serotype pre-post vaccination will be calculated. The average change will then be compared over time for each group and also between healthy and immunosuppressed groups using t-tests. Geometric mean titres of antibody for each serotype will be measured and compared at each follow up interval.

SECONDARY OUTCOMES:
Duration of immunity | 5 years
  Interpretation of Results: Persistance of immunity will be measured over 5 years, as well as the comparison of immunogenicity by immune status.

CONTACTS AND LOCATIONS:
Overall Officials: Raina MacIntyre, Principal Investigator — The University of New South Wales
Locations (1):
- School of Public Health and Community Medicine, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
We would like to share publication(s) that may arise from the study when applicable.

REFERENCES:
- [Result] MacIntyre CR, Shaw P, Mackie FE, Boros C, Marshall H, Barnes M, Seale H, Kennedy SE, Moa A, Hayen A, Chughtai AA, O'Loughlin EV, Stormon M. Immunogenicity and persistence of immunity of a quadrivalent Human Papillomavirus (HPV) vaccine in immunocompromised children. Vaccine. 2016 Aug 5;34(36):4343-50. doi: 10.1016/j.vaccine.2016.06.049. Epub 2016 Jul 9. PMID 27406936
- [Derived] MacIntyre CR, Shaw PJ, Mackie FE, Boros C, Marshall H, Seale H, Kennedy SE, Moa A, Chughtai AA, Trent M, O'Loughlin EV, Stormon M. Long term follow up of persistence of immunity following quadrivalent Human Papillomavirus (HPV) vaccine in immunocompromised children. Vaccine. 2019 Sep 3;37(37):5630-5636. doi: 10.1016/j.vaccine.2019.07.072. Epub 2019 Aug 8. PMID 31402238